CLINICAL TRIAL: NCT06615102
Title: A Prospective Angiotensin II Versus Noradrenaline Trial for Hypotension Management to Reduce Cardiac-surgery Associated Acute Kidney Injury (PAN-AKI)
Brief Title: Reducing Cardiac-surgery Associated Acute Kidney Injury Occurence by Administering Angiotensin II
Acronym: PAN-AKI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UniMS23_0019; 542931418 (Other Grant/Funding Number: German Research Foundation)
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery; Vasoplegia
Keywords: cardiac surgery; acute kidney injury; Angiotensin II
MeSH Terms: conditions — Vasoplegia; Acute Kidney Injury | interventions — Angiotensin II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiotensin II (Experimental): Intravenous infusion through a central line according to the patient's situation. Target medium arterial pressure (MAP): >65mmHg
  Interventions: Drug: Angiotensin II
- Control (Active Comparator): Intravenous infusion through a central line according to the patient's situation. Target medium arterial pressure (MAP): >65mmHg
  Interventions: Drug: Noradrenalin

INTERVENTIONS:
Drug: Angiotensin II — Intravenous infusion through a central line according to the patient's situation. Once an infusion is established, the dose will be titrated as frequently as every 5 minutes, as needed, depending on the patient's condition and target MAP.
  Arms: Angiotensin II
Drug: Noradrenalin — Intravenous infusion through a central line according to the patient's situation. Once an infusion is established, the dose will be titrated as frequently as every 5 minutes, as needed, depending on the patient's condition and target MAP.
  Arms: Control

SUMMARY:
The study intervention focuses on exploring the use of angiotensin II as a primary vasopressor compared to norepinephrine in cardiac surgery patients to investigate whether angiotensin II can reduce the occurrence of moderate/severe acute kidney injury (AKI). Despite its potential, as suggested by trials involving surgical patients, there is currently no human data confirming its effectiveness in preventing moderate/severe AKI in this context. The intervention aims to address this gap by evaluating angiotensin II's impact compared to norepinephrine.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is defined by changes in serum creatinine and/or urine output, according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria. In cardiac surgical patients, the AKI rate is up to 30%, with 1-2% of the patients requiring renal replacement therapy (RRT). Cardiac-surgery associated AKI (CSA-AKI) is associated with increased short- and long-term morbidity and mortality as well as increased hospital costs.

Shock after cardiac surgery is also associated with increased mortality. In the context of cardiac surgery with the use of the cardiopulmonary bypass (CPB), sympathetic nervous system activation and cardiovascular instability are common sequelae. Vasoplegic syndrome is a form of distributive shock that is characterized by low arterial pressure, reduced systemic vascular resistance, and normal or elevated cardiac output. It occurs in 5 to 25% of the patients undergoing cardiac surgery. Patients with vasoplegic shock are at higher risk of organ failure, including AKI, and show increased mortality rates and longer hospital length of stays. Currently, norepinephrine is the established first-line vasopressor for the treatment of vasoplegic shock, but all vasopressors have adverse effects, including myocardial ischemia and arrhythmias. Moreover, in vasoplegic situations, vascular smooth muscle cells may become unresponsive to vasopressors. The underlying mechanisms are complex and include adrenoceptor desensitization, increased nitric oxide (NO) synthesis, activation of adenosine triphosphate-sensitive K+ channels, and vasopressin and corticosteroid deficiency.

Physiologically, the renin-angiotensin-aldosterone system (RAAS) is a hormone system that plays a central role in regulating blood pressure and fluid balance, glomerular filtration rate, and electrolyte levels. Renin, a proteolytic enzyme released by juxtaglomerular cells in response to hypotension, decreases sodium delivery to the distal tubule, activates the sympathetic nervous system, and cleaves angiotensinogen to angiotensin I which is a precursor of the vasoactive angiotensin II. RAAS is regulated by a biofeedback loop. Angiotensin II generation inhibits renin release, whereas renin levels increase when there is insufficient activation of the angiotensin II type 1 receptor. Administration of angiotensin converting enzyme inhibitors (ACEi) and angiotensin II receptor blockers (ARB) and reduced angiotensin II generation cause a corresponding increase in renin levels.

Despite numerous clinical trials using several interventions, a reliable means to prevent AKI remains elusive. Clinical trials focusing on surgical patients suggest that angiotensin II is a potent vasopressor. However, no human data exist whether the application of angiotensin II as a primary vasopressor reduces the occurrence of AKI in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac surgery using cardiopulmonary bypass including coronary artery bypass grafting (CABG) surgery, valve surgery, or combined CABG/valve surgery
2. Elevated risk of AKI as predicted by a score ≥ 1.5 on the following scale:

   1. hemoglobin < 130g/l = 2
   2. creatinine > 1.1 mg/dl = 2
   3. age > 70 years =1.5
   4. New York Heart Association Classification (NYHA) 4 =1.5
   5. Body Mass Index (BMI) > 30 =1.5
3. Adult ≥ 18 years
4. Written informed consent

Exclusion Criteria:

1. Major aortic surgery (aortic arch replacement), transplant surgery, pulmonary thrombendarterectomy, ventricular assist device placement
2. Already receiving inotropic/vasopressor support before surgery
3. Dialysis dependent
4. Pre-existing AKI within the last 30 days
5. Pre-existing chronic kidney injury with an eGFR<20 ml/min/1.73m2
6. Pre-existing significant hypertension (persistent SBP > 180mmHg)
7. Significant pulmonary hypertension (ePSAP > 70mmHg, mPAP > 40mmHg) with right ventricular systolic dysfunction (graded more severe than mild)
8. Hypersensitivity to the active substance or to any of the excipients
9. Pregnancy (a negative pregnancy test for women of childbearing age) or breastfeeding women
10. Persons with any kind of dependency on the investigator or employed by the sponsor/investigator
11. Participation in another interventional trial within the last three months that investigates kidney function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1022 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Rate of AKI KDIGO stage 2 or 3 or death within 72 hours after end of cardiac surgery. | 72 hours after end of surgery

SECONDARY OUTCOMES:
Major Adverse Kidney Events (MAKE90) | 90 after cardiac surgery
  1. MAKE90 (consisting of mortality, dialysis within 90 days, persistent renal dysfunction (defined as serum creatinine ≥ 2x compared to baseline value at day 90)
Severity of Acute Kidney Injury | 72 hours after cardiac surgery
  Number of patients with KDIGO stage 1, KDIGO stage 2 or KDIGO stage 3)
Development or progression of chronic kidney injury | 90 to 120 days after cardiac surgery
  Development or progression of chronic kidney disease based on albuminuria, urine creatinine (and the respective ratio) and serum creatinine or death within 120 days

OTHER OUTCOMES:
Use of additional open-label vasopressors or inotropes | within 72 h after cardiac surgery
Volume of fluid application within the first 72 hours | within 72 h after cardiac surgery
Volume status | within 72 h after cardiac surgery
Time to death | 30 days after cardiac surgery
Time to death | 60 days after cardiac surgery
Time to death | 90 days after cardiac surgery
Days alive and in (index) ICU | From start of intervention until 60 days after cardiac surgery
Days alive and in (index) Hospital | From start of intervention until 60 days after cardiac surgery
Incidence of adverse events (AEs) and serious AEs (SAEs) | From start of intervention until discharge / day 7
Occurence of AKI according to the KDIGO criteria | From start of intervention unto 72 hours after cardiac surgery
Number of patients with persistent renal dysfunction | On day 90 after cardiac surgery
  defined as serum creatinine ≥ 2x compared to baseline value
Number of patients with dialysis renal/replacement therapy | On day 90 after cardiac surgery
Mortality | On day after cardiac surgery
Dose of vasopressors | from start of surgery unto 72 hours after cardiac surgery
Days alive and free of mechanical ventilation until day 60 | From start of intervention unto 60 days after cardiac surgery
Duration of mechanical ventilation | From start of intervention unto discharge from hospital or day seven after cardiac surgery (whatever comes first)
Days alive and free of vasopressors and mechanical ventilation | From start of intervention unto 60 days after cardiac surgery
Number of days alive and free of vasopressors and mechanical ventilation | From start of intervention until 28 days after cardiac surgery
Change in total and individual organ failure scores through 72 hours | Start of intervention and 72 hours after cardiac surgery
  Sequential Organ Failure Assessment (SOFA) score
Duration of renal replacement therapy | From start of intervention unto 90 days after cardiac surgery
Number of patients with renal replacement therapy | Day 90 after cardiac surgery
Creatinine clearance on day one after cardiac surgery | 24 hours after cardiac surgery
Incidence of documented new onset atrial fibrillation | From end of surgery to hospital discharge
Occurrence of transient (< 48 hours) and persistent (≥ 48 hours) AKI | From start of intervention to hospital discharge
Identification and evaluation of biomarkers | From start of intervention to 48 hours after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Principal Investigator — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Medicine and Pain Therapy
Locations (4):
- Germany (4):
  - Deutsches Herzzentrum der Charité, Berlin
  - University Hospital Bonn, Bonn
  - University Medical Center Mainz, Mainz
  - University Hospital Münster, Münster

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be available up to 3 years after original manuscript publication to researchers with methodologically sound proposals approved by the principal investigator.
  Supporting Materials:
Supporting Information: Study Protocol, ICF
Time Frame: Up to 3 years after original manuscript publication
Access Criteria: Available to researchers with methodologically sound proposals approved by the principal investigator.